CLINICAL TRIAL: NCT00604604
Title: An RCT to Evaluate the Effectiveness of Peer (Mother-to-Mother) Support for the Prevention of Postpartum Depression
Brief Title: Postpartum Depression Prevention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Cindy-Lee Dennis, Lawrence S. Bloomberg Faculty of Nursing, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCT-66874; ISRCTN68337727
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2008-01

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control group (usual postpartum care)
- 2 (Experimental): Experimental group (usual postpartum care plus telephone-based support from an experienced mother who has participated in a 4-hour training session)
  Interventions: Behavioral: Peer support

INTERVENTIONS:
Behavioral: Peer support — Mothers allocated to the peer support group had access to all of the standard community postpartum services in addition to having received telephone-based support from a peer volunteer (a mother who has previously experienced, and recovered from, postpartum depression and has participated in a 4-hour training session). Telephone contact with a new mother was initiated within 48 to 72 hours of trial enrolment and then as frequently as the dyad deemed necessary; a minimum of four contacts were required.
  Other Names: Mother-to-mother support
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the effect of peer (mother-to-mother) support on the prevention of postpartum depression among mothers identified as high-risk.

DETAILED DESCRIPTION:
Many new mothers from diverse cultures experience postpartum depression (PPD), a serious form of maternal morbidity with well documented health consequences for the mother, child, and family. While the cause of PPD remains unclear, research consistently demonstrates the importance of psychosocial variables. The purpose of this randomized controlled trial is to evaluate the effect of peer (mother-to-mother) support on the prevention of PPD among mothers identified as high-risk. Public health nurses using the Edinburgh Postnatal Depression Scale (EPDS) screened mothers who were less than 2 weeks postpartum in the regions of Toronto, Peel, Halton, York, Windsor, Sudbury, and Ottawa. Eligible and consenting mothers were randomized to either a control group (usual postpartum care) or experimental group (usual postpartum care plus telephone-based support from an experienced mother who has participated in a 4-hour training session). Diverse study outcomes, including depressive symptomatology and health service utilization, were assessed at 12 and 24 weeks postpartum. The results from this trial will make substantive contributions in six areas: (1) develop the body of knowledge concerning the effectiveness of peer support in the prevention of PPD among at-risk mothers; (2) advance our understanding of the advantages and disadvantages of using peer volunteers as a complementary form of health care; (3) provide an economic evaluation of a peer support intervention; (4) offer a detailed analysis of peer support interactions including supportive functions provided, types of relationships developed, and health benefits perceived; (5) investigate the utility of screening at-risk mothers using the EPDS in general public health nursing practice; and (6) present valuable information regarding PPD among a multicultural Canadian population.

ELIGIBILITY:
Inclusion Criteria:

* live birth
* discharged from hospital
* <2 weeks postpartum
* scored >9 on the EPDS
* availability of a peer volunteer who speaks the potential participant's language

Exclusion Criteria:

* infant not discharged home with mother
* current use of anti-depressant or anti-psychotic medication
* prior self-reported mental illness, including prior PPD, will NOT be an exclusion criterion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2004-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM-IV (SCID-I); Edinburgh Postnatal Depression Scale (EPDS) | 12 weeks postpartum

SECONDARY OUTCOMES:
State Anxiety Inventory (STAI); UCLA Loneliness Scale; Maternal Health Service Utilization and Cost of Care Questionnaire; Peer Support Evaluation Inventory; Peer Volunteer Experience Questionnaire; Peer Volunteer Activity Log | 12 and 24 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Cindy-Lee Dennis, PhD, Principal Investigator — Lawrence S. Bloomberg Faculty of Nursing, University of Toronto
Locations (7):
- Canada (7):
  - Sudbury & District Health Unit, Greater Sudbury, Ontario
  - Peel Health Department, Mississauga, Ontario
  - Halton Region Health Department, Oakville, Ontario
  - Ottawa Public Health, Ottawa, Ontario
  - York Region Health Services, Richmond Hill, Ontario
  - Toronto Public Health, Toronto, Ontario
  - Windsor Essex County Health Unit, Windsor, Ontario